CLINICAL TRIAL: NCT04250740
Title: The Morning Coffee Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Amanda Wright, Ph.D., Associate Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-11-008
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-12

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior | interventions — Coffee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Coffee A (Experimental)
  Interventions: Other: Coffee with butter-1
- Coffee B (Experimental)
  Interventions: Other: Coffee with butter-II
- Coffee C (Experimental)
  Interventions: Other: Coffee with butter-III

INTERVENTIONS:
Other: Coffee with butter-1 — 250 mL brewed black coffee with hazelnut flavouring and 50 g water
  Arms: Coffee A
Other: Coffee with butter-II — 250 mL brewed black coffee with hazelnut flavouring and 50 g unsalted butter-I
  Arms: Coffee B
Other: Coffee with butter-III — 250 mL brewed black coffee with hazelnut flavouring and 50 g unsalted butter-II
  Arms: Coffee C

SUMMARY:
The liking of a breakfast meal has been shown to influence food choice throughout the day. This study will investigate the effects that liking of different coffee beverages has on daily food intake.

DETAILED DESCRIPTION:
This is a postprandial acute meal crossover blinded study in which 30 fasted young healthy women will consume one of 3 butter-rich coffees, in random order, at each of three study sessions separated by at least 4 days. Participants will rate the coffee characteristics and complete paper visual analogue scale ratings of alertness, fatigue, nausea, satiety, and comfort for 180 minutes and consume a pasta lunch meal. A subset of 10 participants will be invited to attend 3 additional study visits where gastric emptying following consumption of each coffee will be assess using gastric ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy women
* 20-35 yrs
* BMI of 18.5-26.1 kg/m2 and waist circumference <88cm
* Non-smoking
* Non to moderate alcohol drinkers
* Regular coffee consumers
* Regularly consumes dairy products
* Pre-menopausal with regular monthly periods
* Stable medication use
* Have not gained or lost significant weight during the past 3 months
* Not pregnant or lactating
* Enjoy and be willing to consume pasta with tomato sauce

Exclusion Criteria:

* Any food sensitivity or intolerance
* Any anaphylactic allergy or gastrointestinal disorder
* History of any major disease or medical condition
* Elite or training athletes
* Three Factor Eating Questionnaire restraint score >16
* Taking any natural health products or dietary supplements, other than a multivitamin, that interfere with fat or caffeine digestion

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We aim to recruit adults with regular menstrual periods, whereby we would include an eligible menstruating participant who identifies as a gender other than female.
Enrollment: 30 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Please indicate how much you liked or disliked the coffee | 30-180 minutes
  Hedonic scale ratings of beverage liking; 9 points from Dislike Extremely to Like Extremely

SECONDARY OUTCOMES:
Please indicate on the line the creaminess of the coffee | 0 - 180 minutes
  Visual analogue scale ratings of product attributes; 0-100 mm from Not Creamy at All to Extremely Creamy
Please indicate on the line how hungry you are | 30 - 180 minutes
  Visual analogue scale ratings of product attributes; 0-100 mm from Not Hungry at All to Extremely Hungry
Lunch meal food intake | 180 minutes
  Weight of food consumed at ad libitum pasta meal

OTHER OUTCOMES:
Gastric emptying | 0, 30, 60, 90, 120, 150, and 180 minutes
  Determined by gastric ultrasound assessment of gastric antrum cross sectional area

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No